CLINICAL TRIAL: NCT06894550
Title: Short-term Exposure to High Altitude in Patients With Asymptomatic Aortic Stenosis
Acronym: ASALT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-00126
Record Dates: First submitted 2025-03-11; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Aortic Stenosis; Altitude
Keywords: Aortic stenosis; High altitude
MeSH Terms: conditions — Aortic Valve Stenosis; Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Prospective, monocentric, three-arm cohort study Group 1: Patients with asymptomatic moderate or severe aortic stenosis Group 2: Patients with aortic stenosis s/p aortic valve replacement Group 3: Age- and sex-matched healthy individuals
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with asymptomatic moderate or severe aortic stenosis (Experimental): Patients with asymptomatic moderate or severe aortic stenosis (moderate or severe aortic stenosis (aortic valve area (AVA) ≤1.5 cm2, NYHA class I, LVEF > 50%, aortic stenosis staging classification Stage 0 or 1)
  Interventions: Behavioral: Participants will be escorted to high altitude and undergo a series of test
- Patients with aortic stenosis s/p aortic valve replacement (Active Comparator): Patients with aortic stenosis s/p aortic valve replacement (aortic stenosis s/p aortic valve replacement within 1 year, NYHA class I , LVEF > 50%, aortic stenosis staging classification Stage 0 or 1)
  Interventions: Behavioral: Participants will be escorted to high altitude and undergo a series of test
- Age- and sex-matched healthy individuals (Active Comparator): Age- and sex-matched healthy individuals ( NYHA class I, LVEF >50%, no evidence of valvular heart disease, age > 65 years)
  Interventions: Behavioral: Participants will be escorted to high altitude and undergo a series of test

INTERVENTIONS:
Behavioral: Participants will be escorted to high altitude and undergo a series of test — Participants will be escorted to high altitude and undergo the following examination both at 540 and 3545m above sea level:
  * 12-lead electrocardiogram
  * Transthoracic echocardiography with measurement of left and right ventricular dimension and function, global longitudinal strain and transvalvular gradient
  * Symptom-limited cardiopulmonary stress exercise test with a ramp protocol with a focused echocardiography for the assessment of cardiac output and transvalvular gradient and blood gas analysis
  * 24 hours wearable rhythm monitoring
  * Blood Work: cardiac biomarkers (Troponin T, CK, CK-MB, NT-pro-BNP), blood gas analysis, Hemoglobin, Hematocrit, Leucocytes, Thrombocytes, Creatinin, eGFR, Sodium, Potassium, ASAT, ALAT, Bilirubin)

SUMMARY:
Aortic stenosis is a common disease with increasing prevalence due to an aging population. Aortic valve replacement is indicated for symptomatic severe aortic stenosis. Leisure activities and tourism at high altitude destinations are popular but may impose a higher risk to patients with aortic stenosis. Pathophysiological considerations led to an expert consensus to avoid high altitude exposure, though there is no robust scientific evidence.

Hence, the objective of this study is to evaluate the safety of high altitude exposure in patients with asymptomatic moderate or severe aortic stenosis by the measurement of surrogate markers for cardiac adverse events such as the decrease in exercise capacity, the assessment of changes in cardiac filling pressures, cardiac dimensions and function, and the evaluation of the incidence of cardiac arrhythmia.

DETAILED DESCRIPTION:
- Hemodynamic changes of high altitude exposure

Atmospheric pressure exponentially decreases with increasing altitude and results in hypobaric hypoxia and arterial hypoxemia. Adaptive mechanisms to high altitude involve the cardiovascular, pulmonary and metabolic system and result in important hemodynamic changes. Acute hypoxia is associated with an increase in cardiac output, heart rate, myocardial contractility, and blood pressure. At the same time, pulmonary vasoconstriction increases pulmonary pressure and right ventricular afterload, while systemic vasodilatation improves peripheral oxygen delivery to the tissues. Hyperventilation furthermore results in respiratory alkalosis and may precipitate premature ventricular complexes and cardiac arrhythmia.

- High altitude exposure in individuals with cardiovascular disease

A range of physiological responses to the high altitude environment challenge the cardiovascular system and potentially increase the risk of adverse cardiovascular events. Pre-existing heart disease can mitigate compensatory mechanisms required for physiological adaption to high altitude. Available evidence is however scarce, which is reflected by the vague clinical recommendations of the European Society of Cardiology and the American Heart Association. Previous evidence suggested that short-term exposure to 3454 meters above sea level was well tolerated in patients with coronary artery disease, stable heart failure and congenital heart disease. There is however no clinical data on the effects of high altitude exposure in patients with valvular heart disease. Expert consensus, based on hemodynamic and pathophysiological considerations, states that patients with symptomatic and/or severe aortic stenosis are prohibited from high altitude exposure/activities.

- Aortic stenosis

Aortic stenosis is the second most prevalent valvular heart disease in the Western World and increases with advancing age. Moderate or severe aortic stenosis was documented in 0.7% of individuals aged ≥65 years in a large-scale community-bases echocardiographic screening program in the United Kingdom, and accounts for more than two thirds of deaths due to degenerative valvular heart disease. The degenerative origin of the disease forecasts an increasing incidence of aortic stenosis in the aging population. An increase in afterload due to aortic valve stenosis leads to an increase in left ventricular pressure and left ventricular wall stress according to the Law of LaPlace. Concentric hypertrophy and an increase in left ventricular mass result in an increased oxygen consumption and a reduction in coronary flow reserve. Upstream cardiac damage may result in mitral regurgitation, left atrial enlargement, pulmonary hypertension, tricuspid regurgitation, and eventually right ventricular dysfunction. The natural history of aortic stenosis is characterized by a long asymptomatic course. Aortic valve replacement is indicated when symptoms such as exercise intolerance, shortness of breath, exertional chest pain or dizziness with syncope develop. Timing of intervention is transitioning from grading of disease according to transvalvular gradients to staging of disease reflecting secondary cardiac damage as a consequence of afterload increase.

- High altitude exposure of individuals with aortic stenosis

Several mechanisms may compromise the short-term adaptation of patients with aortic stenosis to high altitude. An increased oxygen demand of the hypertrophied left ventricle is exacerbated by the hypobaric hypoxia at altitude and may results in myocardial ischemia. This process may be further amplified by an increase in heart rate, and entertain a vicious cycle of myocardial ischemia. At the same time, tachycardia with corresponding increase in cardiac output may aggravate aortic stenosis and precipitate cardiac decompensation. Peripheral vasodilatation may furthermore cause hypotension which is poorly tolerated in aortic stenosis.

- Research question and rationale

Top of Europe/Jungfraujoch located at 3454 meters altitude above sea level is easily accessible by railroad, and visited by more than 1 million tourists every year. Outside of Europe, other tourist hot spots such as Lhasa in Tibet (3658 meters), La Paz in Bolivia (3640 meters), or Cusco in Peru (3399 meters) attract millions of tourists every year. In addition, more than 25 million people worldwide permanently live at an altitude ≥3000 meters. In the absence of robust scientific evidence, even patients with asymptomatic aortic stenosis are discouraged from travelling to high altitude due to hemodynamic considerations. However, data from the Oxvalve registry indicates, that significant valvular heart disease is undiagnosed in 2 out of 3 patients. It can therefore be assumed, that many patients with relevant aortic stenosis travel to high altitude every year without being aware of potential risks.

The goal of the present study is to evaluate the hemodynamic response of patients with asymptomatic moderate or severe aortic stenosis to high altitude, and to assess the safety of high altitude exposure in patients with aortic stenosis. The present study would be the first study to assess the safety of high altitude exposure in patients with aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Moderate or severe aortic stenosis (aortic valve area (AVA) ≤1.5 cm2)
* NYHA class I
* LVEF > 50%
* Aortic stenosis staging classification Stage 0 or 1
* Written informed consent

Group 2:

* Aortic stenosis s/p aortic valve replacement within 1 year
* NYHA class I
* LVEF > 50%
* Aortic stenosis staging classification Stage 0 or 1
* Written informed consent

Group 3:

* NYHA class I
* LVEF >50%
* No evidence of valvular heart disease
* Age > 65 years
* Written informed consent

Exclusion Criteria:

* NYHA class > I (all groups)
* History of cardiac decompensation requiring hospitalization (all groups)
* Uncontrolled arterial hypertension (>180/100 mmHg at rest) (all groups)
* Other Cardiomyopathies w/ normal LVEF (dilatative, hypertrophic, infiltrative CMP) (all groups)
* Signs of exercise-induced ischemia (ST-segment depression > 2 mV), hemodynamic instability (drop in systolic blood pressure > 20 mmHg and systolic blood pressure ≤ 100 mmHg), or ventricular arrhythmias (> 5 beats) during cardiopulmonary stress exercise testing (CPET) at Bern (540 meters) (all groups)
* Chronic obstructive pulmonary disease with a forced expiratory volume in 1 second (FEV1) <60% of the predicted (all groups)
* Known pulmonary hypertension with a pulmonary artery systolic pressure >50 mmHg or high probability of pulmonary hypertension as assessed in TTE (all groups)
* NT-pro BNP levels > 900 pg/ml (all groups)
* Aortic stenosis staging classification > Stage 1 (group 1 and 2)
* History of advanced stages of acute mountain sickness defined as high altitude pulmonary (HAPE) or cerebral (HACE) edema (all groups)
* Transvalvular gradient across the aortic valve ≥60 mmHg, Vmax >5 m/s (group 1)
* Vmax progression ≥0.3 m/s/year (group 1)
* Transvalvular gradient across the aortic valve ≥20 mmHg (group 2)
* Evidence of valvular heart disease or coronary artery disease (group 3)
* History of rhythm disturbances (other than premature ventricular contraction (PVC) (group 3)
* Right ventricular dysfunction, defined as TAPSE < 17 mm, s'DTI < 9 cm/sec (all groups)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety of high altitude exposure in patients with asymptomatic moderate or severe aortic stenosis. Spiroergometry outcome 1 | At end of the investigation at 3545m above sea level, expected to be on average after 3-4 hours
  Decrease in VO2 peak, i.e. VO2-peak @high altitude minus VO2-peak @ low altitude
Safety of high altitude exposure in patients with asymptomatic moderate or severe aortic stenosis. Spiroergometry outcome 2 | At end of the investigation at 3545m above sea level, expected to be on average after 3-4 hours
  Increase in VE/VCO2 slope, i.e. VE/VCO2 slope @high altitude minus VE/VCO2 slope @ low altitude
Safety of high altitude exposure in patients with asymptomatic moderate or severe aortic stenosis. Echocardiography outcome | At end of the investigation at 3545m above sea level, expected to be on average after 3-4 hours
  Increase in left ventricular filling pressure (E/e'), i.e. E/e' @high altitude minus E/e' @ low altitude
Safety of high altitude exposure in patients with asymptomatic moderate or severe aortic stenosis. Rhythmologic outcome | At end of the investigation at 3545m above sea level, expected to be on average after 3-4 hours
  Occurrence of ventricular tachycardia (> 3 beats). Evaluated as presence versus absence.

SECONDARY OUTCOMES:
Symptoms associated with the high altitude exposure | At end of the investigation at 3545m above sea level, expected to be on average after 3-4 hours
  Clinical symptoms of congestive heart failure (NYHA functional class III/IV): Number of patients with newly developed symptoms at high altitude
Laboratory values associated with the high altitude exposure | At end of the investigation at 3545m above sea level, expected to be on average after 3-4 hours
  Increase in NT-proBNP levels. Measurement = NTproBNP @high altitude minus NTproBNP @ low altitude
Arrhythmia associated with the high altitude exposure | At end of the investigation at 3545m above sea level, expected to be on average after 3-4 hours
  Supraventricular or ventricular tachycardia. Number of patients with arrhythmia associated with the high altitude exposure
Hemodynamic effect of the high altitude exposure | At end of the investigation at 3545m above sea level, expected to be on average after 3-4 hours
  Drop in blood pressure (> 20 mmHg). Number of participants with a drop in blood pressure of >20mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, MD, MSc, Study Chair — University Hospital of Bern, Bern, Switzerland
Locations (1):
- University Hospital Inselspital, Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rimoldi SF, Sartori C, Seiler C, Delacretaz E, Mattle HP, Scherrer U, Allemann Y. High-altitude exposure in patients with cardiovascular disease: risk assessment and practical recommendations. Prog Cardiovasc Dis. 2010 May-Jun;52(6):512-24. doi: 10.1016/j.pcad.2010.03.005. PMID 20417345
- [Background] Schmid JP, Nobel D, Brugger N, Novak J, Palau P, Trepp A, Wilhelm M, Saner H. Short-term high altitude exposure at 3454 m is well tolerated in patients with stable heart failure. Eur J Heart Fail. 2015 Feb;17(2):182-6. doi: 10.1002/ejhf.227. Epub 2015 Jan 19. PMID 25597947
- [Background] Schmid JP, Noveanu M, Gaillet R, Hellige G, Wahl A, Saner H. Safety and exercise tolerance of acute high altitude exposure (3454 m) among patients with coronary artery disease. Heart. 2006 Jul;92(7):921-5. doi: 10.1136/hrt.2005.072520. Epub 2005 Dec 9. PMID 16339809